CLINICAL TRIAL: NCT03051048
Title: System Delay and Clinical Outcome Among Chinese Patients With AMI Treated With Reperfusion Therapy (MOODY Study)
Acronym: MOODY
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: NFH20170208
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Coronary Heart Disease
Keywords: Acute Myocardial Infarction
MeSH Terms: conditions — Coronary Disease | interventions — Reperfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The patient received reperfusion therapy between 1999 January 1 and 2009 December 31
  Interventions: Procedure: Reperfusion
- Group 2: The patient received reperfusion therapy between 2010 January 1 and 2016 December 31
  Interventions: Procedure: Reperfusion

INTERVENTIONS:
Procedure: Reperfusion

SUMMARY:
Acute myocardial infarction (AMI) pose a pool clinical outcome to men and women whom treatment was delayed. However, reperfusion time was limited in previous studies. To evaluate the system delay and clinical outcomes among Chinese patients with AMI, consecutive inpatient case prospectively collected from 1999 to 2016. Basic data and innovative evidence will accelerate evidence-based clinical practice and policy making, and improve AMI patients outcomes finally.

DETAILED DESCRIPTION:
AMI is one of the leading causes of mortality and morbidity in public health globally, as well as in China. Remarkable variations of repercussion time and clinical outcome have been noted, however little information is available about how shortened D2B time is incorporated appropriately into routine clinical practice in China. In addition, basic data and evidence about effectiveness of treatment for AMI during long-term recovery is limited. Practical and applied knowledge from large unselected population is needed to guide practice for improvement.

This study will enroll patients with a confirmed diagnosis of AMI consecutively in China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. At 1 month, and 12 month after discharge, participants will return to the clinic for follow up visits. This study will examine system delay that may affect patients recovery after a heart attack. Effective clinic path system, and risk model for AMI patients will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute myocardial infarction according to positive cardiac biomarkers (Troponin I/T, CK-MB or CK≥ local laboratory upper limit of normal values within 24 hours after initial presentation, and at least one of the following two supporting evidence of ischemia (ischemic symptoms occurring within 24 hours before admission or up to 72 hours for STEMI; ECG changes indicative of new ischemia).

Exclusion Criteria:

* Previously enrolled in the similar study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In China, hospitalized patients with acute myocardial infarction will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
30-Day Freedom From Mortality | 30 days
  All-cause death

SECONDARY OUTCOMES:
12-Month Freedom From Major Adverse Cardiac Events (MACE) | 12 months
  Composite of MACE including cardiac death, non-fatal AMI, and clinically driven target vessel revascularization.
Cardiac death | 12 months
  Death that could not be attributed to a noncardiac etiology was considered cardiac death.
Myocardial infarction | 12 months
  Myocardial infarction was diagnosed by electrocardiographic changes and/or a rise and fall of creatine kinase-myocardial band fraction in the presence of ischemic symptoms.
Target vessel revascularization | 12 months
  Target vessel revascularization was defined as repeated revascularization by PCI or surgery of the target vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (23):
- China (23):
  - Changshu First People's Hospital, Changshu, Jiangsu
  - Changzhou Traditional Chinese Medicine Hospital, Changzhou, Jiangsu
  - Jintan People's Hospital, Jintan, Jiangsu
  - Liyang Hospital of TCM, Liyang, Jiangsu
  - Gaochun People's Hospital, Nanjing, Jiangsu
  - Anqing First People's Hospital, Anqing
  - The 123 Hospital of PLA, Bengbu
  - Changzhou Fouth People's Hospital, Changzhou
  - Huaian Second People's Hospital, Huai'an
  - Huainan Eastern Hospital, Huainan
  - Huainan Xinhua Hospital, Huainan
  - Maanshan Shiqiye Hospital, Ma’anshan
  - Muyang Traditional Chinese Medicine Hospital, Muyang
  - Nanjing First Hospital, Nanjing
  - Nanjing Pukou Central Hospital, Nanjing
  - Nnajing 81 Hospital, Nanjing
  - Nnajing Integrated Traditional Chinese and Westem Medicine Hospital, Nanjing
  - Taicang First People's Hospital, Taicang
  - Wuxi Third Hospital, Wuxi
  - Yixin People's Hospital, Wuxi
  - Yixing Traditional Chinese Medicine Hospital, Wuxi
  - Xuncheng Central Hospital, Xuancheng
  - Zhangjiagang First People's Hospital, Zhangjiagang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue X, Kan J, Zhang JJ, Tian N, Ye F, Yang S, Qu H, Chen SL; MOODY trial investigators. Comparison in Prevalence, Predictors, and Clinical Outcome of VSR Versus FWR after Acute Myocardial Infarction: The Prospective, Multicenter Registry MOODY Trial-Heart Rupture Analysis. Cardiovasc Revasc Med. 2019 Dec;20(12):1158-1164. doi: 10.1016/j.carrev.2019.01.023. Epub 2019 Jan 23. PMID 30755362